CLINICAL TRIAL: NCT06036355
Title: THE Exploratory Study on the Biological Function of Dendritic Cells In Vivo Supported by Nicotinamide Mononucleotide (Vital NAD)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH2301-A-03
Record Dates: First submitted 2023-08-15; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Prevention of Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orally take NMN (Vital NAD) combined with DC cell vaccine injection (Experimental): The arm is a combination of two drugs. The first NMN is a precursor of NAD+, which is used orally. DC vaccine is a kind of immune cells expanded in vitro and used by injection.
  Interventions: Drug: Oral NMN combined with DC cell vaccine

INTERVENTIONS:
Drug: Oral NMN combined with DC cell vaccine — The whole intervention cycle was treated with NMN (Vital NAD) 600mg/day for at least 50 days. During this period, the first DC cell injection was given on the 10th day, and then another DC cell injection was given at 2 weeks, 4 weeks and 6 weeks after the first injection.

SUMMARY:
The main purpose of this study is to explore the PK/PD changes of NMN and DC cells after oral NMN combined with DC cells injection in patients after tumor surgery, and evaluate the biological age of adults, TCR diversity, SiRT1 expression level, SF-36 quality of life, OS, antigen specific immune response (TAA), cytokines and so on. In this study, 20 postoperative tumor patients who meet the entry and excretion criteria were recruited to explore the clinical potential of NMN combined with DC cell vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-80 years old, weight ≥ 40kg.
* 2. Patients with malignant solid tumors diagnosed by histology or cytology, who underwent radical resection and completed standard postoperative adjuvant therapy.
* 3. Estimated survival time ≥ 6 months.
* 4. ECOG score 0-1.
* 5. Adequate venous channels, there is no contraindication for peripheral blood monocyte collection.
* 6. Good function of organs and bone marrow.

Exclusion Criteria:

* 1. Diabetes.
* 2. Premenopausal or menopause <1 year.
* 3. Persons who have received hormone replacement therapy within the past 6 months.
* 4. Persons who take vitamin B supplementation and are not willing to discontinue supplementation for 3 weeks before and during the entire study period.
* 5. Unstable weight (>3% change during the last 2 months before entering the study).
* 6. Significant organ system dysfunction or disease.
* 7. Polycystic ovary syndrome.
* 8. Major psychiatric illness.
* 9. Use of medications known to affect study outcome measures (e.g., steroid) or increase the risk of study procedures (e.g., anticoagulants) that cannot be temporarily discontinued for the study.
* 10. Metal implants.
* 11. Persons who consume >14 units of alcohol per week.
* 12. Unable or unwilling to follow the study protocol or who, for any reason, is considered an inappropriate candidate for the study by the research team.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of double antibodies in peripheral blood | Up to 3 months
Concentration of NMN (nicotinamide mononucleotide) in peripheral blood | Up to 3 months
Peripheral blood NAD+ | Up to 3 months
Cytokines (IL6, TNF- goat, INF- γ, IL-4, IL-10) | Up to 3 months
T cell depletion index (PD1/Tim-3/lag3) | Up to 3 months
T cell activation index CD107 | Up to 3 months
T cell and NK cell function index (INF- γ) and granzyme | Up to 3 months
High quality Survival benefit Endpoint (DFS) | Up to 15 years
  DFS refers to the time from the beginning of treatment to the recurrence of the disease or the death of the patient. Patients need to be followed up regularly to keep records.
Survival benefit (OS) | Up to 15 years
  OS refers to the time from the beginning of randomization to death (for any reason). Patients need to be followed up regularly to keep records.
Distant Metastasis-Free Survival (DMFS) | Up to 15 years
  Metastasis-free survival time. Patients need to be followed up regularly to keep records.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR